CLINICAL TRIAL: NCT02169947
Title: Weight Loss and Maintenance for Rural, African American Communities of Faith (The WORD)
Acronym: WORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 134125; 2P20MD002329-06 (NIH)
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Maintenance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight loss core (Active Comparator): Participants will receive a culturally adapted version of the Diabetes Prevention Program core (16 session) program.
  Interventions: Behavioral: Weight loss core
- Weight loss core plus maintenance (Experimental): Participants will receive a culturally adapted version of the Diabetes Prevention Program core (16 session) program PLUS 12 maintenance sessions.
  Interventions: Behavioral: Weight loss core; Behavioral: Weight loss core plus maintenance

INTERVENTIONS:
Behavioral: Weight loss core — The weight loss core is a culturally adapted version of the Diabetes Prevention Program core 16 week session program.
Behavioral: Weight loss core plus maintenance — The intervention is a culturally adapted version of the Diabetes Prevention Program core 16 sessions plus 12 maintenance sessions.
  Arms: Weight loss core plus maintenance

SUMMARY:
The WORD (Wholeness, Oneness, Righteousness, Deliverance) is a faith-based weight loss study in rural, African American adults of faith. The study will see whether a weight loss + maintenance intervention will cause participants to maintain their weight better than a weight loss only intervention.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Aged 18 and older
* Have a BMI ) > 25 kg/m²
* Associated with a participating church through membership or participation in a church activity
* Free of medical problems that might contraindicated participation in a behavioral weight reduction program containing an exercise component
* Individuals taking sulfonylureas who have a letter from their doctor supporting their participation in the study will be considered eligible

Exclusion Criteria

* Not had a heart attack or stroke in the past 6 months
* Not currently on medication that might affect weight loss or require medical monitoring (i.e. insulin)
* Not pregnant, not pregnant in the previous six months, or lactating
* Not enrolled in another weight reduction program
* Agree to complete the program assigned to them
* Never had weight loss surgery
* Not have lost more than 10% body weight in the previous 6 months
* Not have a clinically significant medical condition likely to impact weight or any condition that makes it unlikely the participant would be available to follow the protocol for 18 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Change in weight from 6 months to 18 months | Change from 6 months to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeary, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States